CLINICAL TRIAL: NCT01859481
Title: A Multicentre, Dose Optimisation Study to Assess the Consistency of Efficacy of Eletriptan for the Treatment of Migraine (With and Without Aura)
Brief Title: Eletriptan Provides Consistent Migraine Relief: Results Of A Within-Patient Multiple-Dose Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1601015
Record Dates: First submitted 2013-05-13; First posted 2013-05-22 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Migraine Without Aura; Migraine With Aura
MeSH Terms: conditions — Migraine without Aura; Migraine with Aura | interventions — eletriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Eletriptan HBr 40 mg (Experimental)
  Interventions: Drug: Eletriptan HBr 40 mg
- Eletriptan HBr 80 mg (Experimental)
  Interventions: Drug: Eletriptan HBr 80 mg

INTERVENTIONS:
Drug: Placebo — All subjects will receive open label eletriptan 40 mg per attack for the first three attacks in the phase 1 of the study. For the next 4 attacks subjects will be assigned to either eletriptan 40 mg or 80 mg group based on the response in the phase 1 portion of the study. In phase II, in each group subjects will receive eletriptan 40 mg or 80 mg for 3 attacks and placebo for 1 attack. In each group double-blind placebo will be inserted at random.
  Arms: Placebo
Drug: Eletriptan HBr 40 mg — All subjects will receive open label eletriptan 40 mg per attack for the first three attacks in the phase 1 of the study. For the next 4 attacks subjects will be assigned to either eletriptan 40 mg or 80 mg group based on the response in the phase 1 portion of the study. In phase II, in each group subjects will receive eletriptan 40 mg or 80 mg for 3 attacks and placebo for 1 attack. In each group double-blind placebo will be inserted at random.
  Arms: Eletriptan HBr 40 mg
Drug: Eletriptan HBr 80 mg — All subjects will receive open label eletriptan 40 mg per attack for the first three attacks in the phase 1 of the study. For the next 4 attacks subjects will be assigned to either eletriptan 40 mg or 80 mg group based on the response in the phase 1 portion of the study. In phase II, in each group subjects will receive eletriptan 40 mg or 80 mg for 3 attacks and placebo for 1 attack. In each group double-blind placebo will be inserted at random.
  Arms: Eletriptan HBr 80 mg

SUMMARY:
Evaluation of headache response at 2 hours for active treated attacks for increasing dose.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects in good general health, aged 18 to 65 years.
* Subjects should meet IHS diagnostic criteria for migraine with or without aura.
* Based on past history, subjects should expect to suffer at least one acute attack of migraine with or without aura, each 6 weeks

Exclusion Criteria:

* Known coronary-artery disease, clinically significant arrhythmia, heart failure, or uncontrolled hypertension.
* Pregnant or lactating women.
* Clinically significant electrocardiogram abnormalities at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 971 (Actual)
Dates: Start 2000-03; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Consistency of headache response (3 responses out of 3 active treated attacks) . Headache response was defined as migraine headache pain of moderate or severe intensity pre dose becoming basent or mild within 2 hours post dose. | 24 weeks

SECONDARY OUTCOMES:
Consistency of headache response (2 responses out of 3 active treated attacks). Headache response was defined as migraine headache pain of moderate or severe intensity pre dose becoming basent or mild within 2 hours post dose. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (147):
- Belgium (5):
  - Eeuwfeestkliniek, Antwerp
  - A.Z. Sint Jan, Bruges
  - Cliniques Universitaires St Luc, Brussels
  - C.H.U. de Charleroi, Charleroi
  - Hopital de La Citadelle, Liège
- Czechia (4):
  - Faculty Hospital U Svety Anny, Brno
  - Neurologika Klinika F.N., Hradec Králové
  - Pain Centrum, Prague
  - 1St Medical Faculty of the Charles University, Prague
- Denmark (5):
  - Arhus Kommunehospital, Arhus C
  - Kas Glostrup, Glostrup Municipality
  - Korsgaard, Anne G. (Private Practice), Odense C
  - Asbjorn Ziebel, Roskilde
  - Peter Staehr, Ølstykke
- France (24):
  - Hopital de Rangueil, Toulouse, Cedex 04
  - Veyrie-Courtade, Toulouse, Tououse
  - C.H.U.R Bretonneau, Tours, Tours
  - Kubler Altkirch, Altkirch
  - Marcombes Angouleme, Angoulême
  - Houdart Anzin, Anzin
  - Groupe Pellegrin Tripode, Bordeaux
  - Siboni Carcassonne, Carcassonne
  - Hopital Louis Mourier, Colombes
  - Cormier Laval, Laval
  - Hopital Salengro, Lille
  - Hopital Louis Pradel, Lyon
  - Hopital Pasteur, Nice
  - Private Practice, Orléans
  - Delfiner Paris, Paris
  - Hopital Lariboisiere, Paris
  - Hopital Cochin, Paris Codex 14
  - Vaunaize Reims (Ds For Oc), Reims
  - Vaunaize Reims, Reims
  - Hopital Charles Nicolle, Rouen
  - Hospital Bellevue, Saint-Etienne
  - Bouchacourt Toulon, Toulon
  - Lemarquis Toulon, Toulon
  - Mick Voiron, Voiron
- Germany (9):
  - Private Practice, Berlin
  - Private Practice (Guenther Schumann), Bochum
  - Private Practice, Bochum
  - Private Practice, Eckernförde
  - Private Practice, Göttingen
  - Private Practice, Hamburg
  - Private Practice, Oldenburg
  - Fachklinik Fuer Neurologie Dietenbronn Gmbh, Schwendi
  - Private Practice (Dr. Renate Kreyer), Stade
- Greece (3):
  - Neurology Clinic of Chania, Soúda, Chania,crete
  - General Athens State Hospital, Athens
  - Saint Dimitrios Hospital, Thessaloniki
- Hungary (7):
  - Peterfy Teaching Hospital, Budapest
  - Semmelweis University, Budapest
  - Szent-Imre Hospital, Budapest
  - Jahn Ferenc Hospital, Budapest
  - Uzsoki Hospital, Budapest
  - University of Debrecen, Medical and Health Science Centre, Medical School, Debrecen
  - Kenezy County Hospital, Debrecen
- Italy (18):
  - Universita Degli Studi Di Modena-Policlinico Dipartimento Di Medicina Interna, Modena, Emilia-Romagna
  - Fondazione Istituto Neurologico Casimiro Mondino Istituto Di Ricovero E Cura A Carattere Scientifico, Pavia, Lombardy
  - Universita' Di Bologna, Bologna
  - Poliambulatorio Salus, Brescia
  - Universita' Degli Studi Di Cagliari - Presidio Osp.S.Giovanni Di Dio, Cagliari
  - Azienda Vittorio Emanuele, Catania
  - Clinica Neurologica, L'aquila-coppito
  - Policlinico Universitario, Messina
  - Centro Cefalee Irccs "C. Besta", Milan
  - Universita Di Padova, Padua
  - Centro Cefalee, Parma
  - Clinica Neurologica, Universita Di Perugia, Perugia
  - Centro Cefalee - Neuromed, Pozzilli (isernia)
  - Ospedale S. Eugenio, Roma
  - Centro Cefalee, Torino
  - Ospedale Regionale Torrette, Torrette DI Ancona (AN)
  - Ospedale Maggiore, Trieste
  - Ospedale S. Bortolo, Vicenza
- Netherlands (12):
  - Bosch Medicentrum (Locatie Willem Alexander Ziekenhuis), 's-Hertogenbosch
  - Sint Lucas Andreas Ziekenhuis (Location: St.Lucas), Amsterdam
  - Gelre Ziekenhuis (Location: Lukas), Apeldoorn
  - Ziekenhuis Gooi-Noord, Blaricum
  - Ignatius Ziekenhuis Breda, Breda
  - Gelderse Vallei Ziekenhuis, Ede
  - Scheperziekenhuis, Emmen
  - Atrium Heerlen, Heerlen
  - St. Streekziekenhuis Midden Twente, Hengelo (OV)
  - Ikazia Ziekenhuis, Rotterdam
  - Sint Elisabeth Ziekenhuis, Venray
  - Lage Land Ziekenhuis, Zoetermeer
- Norway (3):
  - Sentralsykehuset I Akershus, Nordbyhagen
  - Volvat Medisinske Senter, Oslo
  - Strandquist, Dr. Stein Bror, Tønsberg
- Portugal (3):
  - Hospital Garcia Da Orta, Almada
  - Centro Hospitalar de Coimbra, Coimbra
  - Hospital S.Joao, Porto
- Spain (20):
  - Consorci Hospitalari Del Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario de Puerto Real, Puerto Real, Cadiz
  - Fundacion Hospital Alcorcon, Alcorcón, Madrid
  - Hospital de Galdakao, Galdakao, Vizcaya
  - Hospital Torrecardenas, Almería
  - Hospital Del Sagrado Corazon, Barcelona
  - Hospital General Universitari Vall D�Hebron, Barcelona
  - Hospital General Yag�, Burgos
  - Hospital Nuestra SE�Ra de Alarcos, Ciudad Real
  - Hospital Na Sa de Aranzazu, Donostia / San Sebastian
  - Hospital Ciudad de Jaen, Jaén
  - Hospital Universitari de Lleida Arnau de Vilanova, Lleida
  - Hospital Ramon Y Cajal, Madrid
  - Hospital Universitario San Carlos, Madrid
  - Hospital Virgen de La Victoria, Málaga
  - Hospital General Universitario J. M. Morales Meseguer, Murcia
  - Hospital General de Asturias, Oviedo
  - Hospital Nuestra SE�Ra de Valme, Seville
  - Hospital Clinico Universitario La Fe, Valencia
  - Hospital General Universitario, Valencia
- Sweden (24):
  - Fritsla Vardcentral, Fritsla
  - Migranklinik-Goeteborg, Gothenburg
  - Lanssjukhuset Halmstad, Halmstad
  - Viktoriakliniken, Halmstad
  - Neurologsektionen, Lasarettet, Helsingborg
  - Neuro Kliniken, Helsingborg, Helsingborg
  - Sjocrona Vardcentral, Höganäs
  - Huddinge Universitetssjukhus, Huddinge
  - Kistahalsan Ab, Kista
  - Lund Lakarmottagningen, Lund
  - Medicin Kliniken, Universitetssjukhuset, Lund
  - Lakargruppen Gustaf Adolf, Malmo
  - Previa Ab Sigtunahalsan, Märsta
  - Oxelohalsan, Oxelösund
  - Bankhalsan, Stockholm
  - Lakarhuset Odenplan, Stockholm
  - Ostermalmshalsan, Stockholm
  - St Gorans Sjukhus, Stockholm
  - Tyresohalsan Huslakare Ab (Ds For Oc), Tyreso
  - Tyresohalsan Huslakare Ab, Tyreso
  - Kronobergskliniken, Vaxjo
  - Centrallasarettet, Västerås
  - Vasterviks Sjukhus, Västervik
  - Novakliniken, Ystad
- Turkey (Türkiye) (2):
  - Cukurova University Medical Faculty, Adana
  - Karadeniz Technical University Medical Faculty, Trabzon
- Country not given (8):
  - Ahepa University Hospital
  - Foretagshalsovarden Linden
  - Huslakargruppen
  - Limhamns Lakargrupp, Tarnan
  - Medicinskt Centrum
  - Sentralsjukehuset I Hedmark
  - Sint Anna Ziekenhuis
  - Vardcentralen

REFERENCES:
- [Derived] Almas M, Tepper SJ, Landy S, Schweizer E, Ramos E. Consistency of eletriptan in treating migraine: Results of a randomized, within-patient multiple-dose study. Cephalalgia. 2014 Feb;34(2):126-35. doi: 10.1177/0333102413500726. Epub 2013 Aug 14. PMID 23946318
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1601015&StudyName=Eletriptan%20Provides%20Consistent%20Migraine%20Relief%3A%20Results%20Of%20A%20Within-Patient%20Multiple-Dose%20Study